CLINICAL TRIAL: NCT07078890
Title: Effect of Bone Augmentation Simultaneous to Implant Removal on the Prognosis of Reimplantation at the Same Site
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Collaborators: Hospital of Stomatology, Wuhan University (Other); Shanghai Stomotological Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-025
Record Dates: First submitted 2025-07-13; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Implant Failure; Bone Augmentation; Prognosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone augmentation simultaneous to implant removal (Experimental): Placement of bone substitutes in the socket simultaneous to implant removal, and reimplantation is performed after 6 months of healing.
  Interventions: Procedure: bone augmentation simultaneous to implant removal
- Natural healing after implant removal (No Intervention)

INTERVENTIONS:
Procedure: bone augmentation simultaneous to implant removal — Placement of bone substitutes in the socket simultaneous to implant removal, and reimplantation is performed after 6 months of healing.
  Arms: Bone augmentation simultaneous to implant removal

SUMMARY:
The aim of this study was to investigate the effect of bone augmentation simultaneous to implant removal on the prognosis of reimplantation at the same sites, providing recommendations for management strategies after failed implant removal.

DETAILED DESCRIPTION:
The study aims to compare the radiographic and clinical indicators between bone augmentation simultaneous to implant removal and natural healing after implant removal, thus evaluate the effect on the prognosis of reimplantation. At the same time, patients with implant failure were also retrospectively collected to investigate the factors influencing the prognosis of bone healing and reimplantation after implant failure.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age greater than 18 years 2. Implant failure requiring removal 3. Plan to reimplant in the same site 4. Periodontal health, or stabilized periodontitis after treatment

Exclusion Criteria:

* 1. Uncontrolled metabolic diseases 2. Taking medications that have an effect on bone metabolism 3. The implant has detached at the time of consultation 4. Do not consent to reimplant in the same site 5. Unwillingness to participate in the follow-up of this study 6. Other conditions that do not qualify for implant therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Ridge Height (RH) | Before implant removal and 6 months after implant removal
  Two reference lines were established for the radiological analysis: the longitudinal axis of the implant and a line perpendicular to this axis and tangential to a reference point (sinus floor in the maxilla and mandibular base in the mandible).Ridge height (RH) in mm, defined as the distance between the tangential reference line and the most coronal point of the bone crest, assessed buccal (B-RH) and lingual (L-RH).

SECONDARY OUTCOMES:
Ridge Width (RW) | Before implant removal and 6 months after implant removal
  Two reference lines were established for the radiological analysis: the longitudinal axis of the implant and a line perpendicular to this axis and tangential to a reference point (sinus floor in the maxilla and mandibular base in the mandible).Ridge width (RW) in mm, recorded at 1, 3, and 5 mm from the bone crest. In the event of discrepancy between the buccal and lingual bone crests, the most apical one was chosen as reference.
Bone Plate Thickness (BPT) | Before implant removal and 6 months after implant removal
  Two reference lines were established for the radiological analysis: the longitudinal axis of the implant and a line perpendicular to this axis and tangential to a reference point (sinus floor in the maxilla and mandibular base in the mandible).Bone plate thickness (BPT) in mm, assessed at 1, 3, 5, and 7 mm below the crest and measured buccal and lingual.
Bone Mineral Density(BMD) | 6 months after implant removal
  Bone density in the socket 6 months after implant removal
Inserting Torque(IT) | Replantation surgery
Implant Survival Rate(SVR) | 6 months and 12 months after restoration
Probing Depth | 6 months and 12 months after restoration
Bleeding On Probing（BOP） | 6 months and 12 months after restoration
Marginal Bone Loss(MBL) | 6 months and 12 months after restoration
  MBL was defined as the linear distance (in mm) measured at both the proximal and distal mesial planes from the most coronal point of the surrounding bone to the cervical plane of the implant.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Hospital of Stomatology, Wuhan University, Wuhan, Hubei
  - The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Shanghai Stomatological Hospital, Shanghai